CLINICAL TRIAL: NCT00217048
Title: Effect of Oral Yohimbine on Colonic Transit: Randomized, Placebo-Controlled Trial
Brief Title: Effect of Yohimbine on Colon Transit
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 275-05
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Yohimbine

INTERVENTIONS:
Drug: Yohimbine, oral

SUMMARY:
This study is being done to learn if yohimbine, a naturally occurring drug, affects the speed at which food travels through the stomach, intestines and colon, and if yohimbine affects the amount of liquid you can drink in a short period of time. Understanding how yohimbine works on the gut may help develop new treatments for patients with constipation. Yohimbine has been approved by the Food and Drug Administration (FDA) for routine clinical use, however, its use as proposed in this study is considered investigational.

ELIGIBILITY:
* Healthy male or non-pregnant, non-breastfeeding female volunteers, -18-65 years old;
* Able to provide written informed consent before participating in the study;
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Colonic transit

SECONDARY OUTCOMES:
Small bowel transit time
Gastric emptying time
Maximum tolerated volume ingested during satiation testing
Average stools per day
Stool consistency

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MBBS, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States